CLINICAL TRIAL: NCT00809965
Title: A Randomized, Double-Blind, Placebo-Controlled, Event-Driven Multicenter Study to Evaluate the Efficacy and Safety of Rivaroxaban in Subjects With a Recent Acute Coronary Syndrome
Brief Title: An Efficacy and Safety Study for Rivaroxaban in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014710; RIVAROXACS3001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-08

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Myocardial Ischemia; Unstable Angina
Keywords: Rivaroxaban; Acute Coronary Syndrome; ACS; Aspirin; Thienopyridine; Unstable Angina; Myocardial Infarction; Anticoagulation; Clopidogrel (Plavix)
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Myocardial Ischemia; Angina, Unstable | interventions — Rivaroxaban; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rivaroxaban 2.5 mg bid (Experimental): One 2.5 mg rivaroxaban tablet twice daily for up to 6 months
  Interventions: Drug: Rivaroxaban 2.5 mg; Drug: Standard of care
- Rivaroxaban 5 mg bid (Experimental): One 5 mg rivaroxaban tablet twice daily for up to 6 months
  Interventions: Drug: Rivaroxaban 5 mg; Drug: Standard of care
- Placebo (Placebo Comparator): One placebo tablet twice daily for up to 6 months
  Interventions: Drug: Placebo; Drug: Standard of care

INTERVENTIONS:
Drug: Rivaroxaban 2.5 mg — One tablet twice daily
  Arms: Rivaroxaban 2.5 mg bid
Drug: Rivaroxaban 5 mg — One tablet twice daily
  Arms: Rivaroxaban 5 mg bid
Drug: Placebo — One placebo tablet twice daily
  Arms: Placebo
Drug: Standard of care

SUMMARY:
The purpose of this study is to determine whether rivaroxaban in addition to standard care reduces the risk of the composite of cardiovascular death, myocardial infarction, or stroke in patients with a recent acute coronary syndrome compared with placebo.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is a serious and life threatening condition. Following an acute coronary syndrome event patients are at risk of important additional clinical events such as death, myocardial infarction, and stroke. Six months after patients present with an index event of ST-segment myocardial infarction, approximately 15% will either have died or had another episode of myocardial ischemia, and a similar situation exists for non-ST-segment elevation myocardial infarction/unstable angina patients. This randomized; double-blind; placebo controlled study will evaluate the efficacy and safety of rivaroxaban in addition to standard care in patients with a recent ACS. Patients will be given rivaroxaban (2.5 mg twice daily or 5 mg twice daily) or placebo (twice daily) in addition to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be currently receiving aspirin therapy alone or in combination with a thienopyridine per national or local dosing recommendation
* Have been hospitalized for symptoms suggestive of acute coronary syndrome that lasted at least 10 minutes at rest and occurred 48 hours or less before going to the hospital

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, contraindicates anticoagulant therapy or would have an unacceptable risk of bleeding
* Need for continued anticoagulant therapy
* Significant renal impairment or known significant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15526 (Actual)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (556):
- United States (73):
  - Birmingham, Alabama
  - Geneva, Alabama
  - Mobile, Alabama
  - Anaheim, California
  - Burbank, California
  - Los Angeles, California
  - Mission Hills, California
  - San Diego, California
  - Aurora, Colorado
  - Littleton, Colorado
  - Jacksonville, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - St. Petersburg, Florida
  - Columbus, Georgia
  - Rome, Georgia
  - Aurora, Illinois
  - Indianapolis, Indiana
  - Merrillville, Indiana
  - Munster, Indiana
  - Valparaiso, Indiana
  - Overland Park, Kansas
  - Wichita, Kansas
  - Lacombe, Louisiana
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Flint, Michigan
  - Grand Blanc, Michigan
  - Grand Rapids, Michigan
  - Kalamazoo, Michigan
  - Mount Clemens, Michigan
  - Petoskey, Michigan
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Kalispell, Montana
  - Bridgewater, New Jersey
  - Linden, New Jersey
  - Buffalo, New York
  - Cortlandt Manor, New York
  - Saratoga Springs, New York
  - Stony Brook, New York
  - Syracuse, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Fairview Park, Ohio
  - Bartlesville, Oklahoma
  - Oklahoma City, Oklahoma
  - Doylestown, Pennsylvania
  - Langhorne, Pennsylvania
  - Ridley Park, Pennsylvania
  - Sayre, Pennsylvania
  - West Chester, Pennsylvania
  - York, Pennsylvania
  - Greenville, South Carolina
  - Johnson City, Tennessee
  - Memphis, Tennessee
  - Amarillo, Texas
  - Lubbock, Texas
  - Odessa, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Danville, Virginia
  - Roanoke, Virginia
  - Spokane, Washington
  - Wausau, Wisconsin
- Argentina (13):
  - Buenos Aires
  - Corrientes
  - Córdoba
  - Junín
  - La Plata
  - Mar del Plata
  - Morón
  - Resistencia
  - Rosario
  - Salta
  - San Luis
  - San Miguel de Tucumán
  - Santa Fe
- Australia (15):
  - Bedford Park
  - Chermside
  - Coffs Harbour South
  - Douglas
  - Epping
  - Fremantle
  - Heidelberg
  - Herston
  - Launceston
  - Milton
  - Newcastle
  - Parkville
  - Perth
  - Southport
  - Woolloongabba
- Belgium (8):
  - Bonheiden
  - Brussels
  - Eupen
  - Genk
  - Huy
  - Leuven
  - Mol
  - Tienen
- Brazil (12):
  - Belo Horizonte
  - Blumenau
  - Campina Grande do Sul
  - Campinas
  - Curitiba
  - Porto Alegre
  - Recife
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - São José do Rio Preto
  - São Paulo
- Bulgaria (11):
  - Burgas
  - Dimitrovgrad
  - Haskovo
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Rousse
  - Sevlievo
  - Sofia
  - Varna
  - Veliko Tarnovo
- Canada (19):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Maple Ridge, British Columbia
  - Victoria, British Columbia
  - St. John's, Newfoundland and Labrador
  - Greater Sudbury, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Granby, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Charles-Borromée, Quebec
  - Saint-Georges, Quebec
  - Sherbrooke, Quebec
  - Ste-Foy, Quebec
  - North Battleford, Saskatchewan
  - Laval
- Chile (12):
  - Antofagasta
  - Chile
  - Osorno X Región
  - Punta Arenas
  - San Bernardo
  - Santiago
  - Santiago Rm
  - Talcahuano
  - Temuco
  - Valdivia X Región
  - Victoria
  - Viña del Mar
- China (13):
  - Beijing
  - Beijing Prc
  - Changsha
  - Daqing
  - Guangzhou
  - Hangzhou
  - Harbin
  - Jinan
  - Nanjing
  - Shanghai
  - Shenyang
  - Tianjin
  - Xi'an
- Colombia (8):
  - Armenia
  - Barranquilla
  - Bogotá Dc
  - Cali Valle Del Cauca
  - Envigado
  - Manizales
  - Medellín
  - Santander
- Croatia (3):
  - Rijeka
  - Slavonski Brod
  - Suska 6
- Czechia (18):
  - Benešov nad Černou
  - Brno
  - České Budějovice
  - Český Krumlov
  - Hradec Králové
  - Kolín
  - Kroměříž
  - Litomyšl
  - Náchod
  - Pardubice
  - Plzeò 1
  - Poruba
  - Prague
  - Praha 10 N/A
  - Slaný
  - Teplice
  - Ústí nad Labem
  - Znojmo
- Denmark (7):
  - Aalborg
  - Copenhagen
  - Esbjerg
  - Holbæk
  - Horsens
  - Kolding
  - Odense
- Egypt (4):
  - Alexandria
  - Cairo
  - Ismailia
  - Menofeya
- France (12):
  - Besançon
  - Cannes
  - Chambray-lès-Tours
  - Chartres
  - Créteil
  - Dijon
  - Haguenau
  - Lagny
  - Marseille
  - Montfermeil
  - Paris
  - Poitiers
- Germany (23):
  - Bad Friedrichshall
  - Berlin
  - Bonn
  - Dresden
  - Essen
  - Esslingen am Neckar
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Göttingen
  - Greifswald
  - Halle
  - Hamburg
  - Hanover
  - Heidelberg
  - Kiel
  - Leipzig
  - Limburg
  - Lübeck
  - Magdeburg
  - Mannheim
  - Weiden
  - Wermsdorf
  - Witten
- Greece (4):
  - Athens
  - Larissa
  - Rhodes
  - Thessalonikis
- Hungary (9):
  - Budapest
  - Debrecen
  - Győr
  - Kecskemét
  - Komárom
  - Miskolc
  - Szolnok
  - Szombathely
  - Zalaegerszeg
- India (29):
  - Ahmedabad
  - Allahabād
  - Bangalore
  - Chandigarh
  - Chennai
  - Coimbatore
  - Ernākulam
  - Gandhinagar Guiarat
  - Gūrgaon
  - Hyderabad
  - Jaipur
  - Karamsad
  - Kochi
  - Kolkata
  - Lucknow Gpo
  - Ludhiana
  - Madurai
  - Mangalore
  - Mumbai
  - Mysore
  - Nagpur
  - Nashik
  - New Delhi
  - Pune
  - Surat
  - Trissur
  - Trivandrum
  - Vadodara
  - Vijayawada
- Israel (10):
  - Afula
  - Hadera
  - Haifa
  - Jerusalem
  - Nahariya
  - Petah Tikva
  - Rehovot
  - Safed
  - Tel Aviv
  - Tiberias
- Japan (38):
  - Anan
  - Fukui
  - Fukuoka
  - Fukuyama
  - Gifu
  - Higashiosaka
  - Kagoshima
  - Kanazawa
  - Kasuga
  - Kawachi-Nagano
  - Kawasaki
  - Kisarazu
  - Kobe
  - Kumamoto
  - Kuwana
  - Maebashi-City Gunma
  - Matsudo
  - Matsumoto
  - Matsuyama-City Ehime
  - Miyazaki-Gun
  - Nagano
  - Nagasaki
  - Nagoya
  - Namegata
  - Nankoku
  - Nishinomiya
  - Okayama
  - Osaka
  - Sakaidechō
  - Sakura-Shi
  - Suwa
  - Tokushima
  - Tokyo
  - Toyama
  - Urasoe
  - Yamaguchi
  - Yokohama
  - Yonago-Shi
- Latvia (3):
  - Daugavpils
  - Liepāja
  - Riga
- Lithuania (5):
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
  - Vilnius Lt
- Malaysia (5):
  - Johor Bahru
  - Kelantan
  - Kota Samarahan
  - Kuala Lumpur
  - Selayang Baru Utara
- Mexico (13):
  - Aguascalientes
  - Cd. Juarez
  - Culiacán
  - Guadalajara
  - León
  - Mexico City
  - México
  - Monterrey
  - Querétaro
  - San Luis Potosí City
  - Sinaloa
  - Veracruz
  - Zapopan
- Morocco (3):
  - Marrakesh
  - Meknes
  - Rabat
- Netherlands (14):
  - Amsterdam
  - Arnhem
  - Delft
  - Eindhoven
  - Gorinchem
  - Gouda
  - Haarlem
  - Harderwijk
  - Hengelo Ov
  - Nieuwegein
  - Nijmegen
  - Sittard
  - The Hague
  - Vlaardingen
- New Zealand (6):
  - Auckland
  - Dunedin
  - Hamilton
  - Lower Hutt
  - Nelson
  - New Plymouth
- Philippines (3):
  - Iloilo City
  - Marikina City
  - Quezon City
- Poland (26):
  - Będzin
  - Bialystok
  - Bielsko-Biala
  - Bydgoszcz
  - Bytom
  - Dąbrowa Górnicza
  - Gdynia
  - Gorlice
  - Katowice
  - Katowice-Ochojec
  - Koszalin
  - Krakow
  - Kutno
  - Lodz
  - Nowy Targ
  - Opole
  - Poznan
  - Płock
  - Ruda Śląska
  - Starogard Gdanski Nap
  - Szczecin
  - Torun
  - Warsaw
  - Wroclaw
  - Włocławek
  - Zamość
- Portugal (9):
  - Aveiro
  - Braga
  - Coimbra
  - Faro
  - Leiria
  - Lisbon
  - Penafiel
  - Porto
  - Vila Nova de Gaia
- Romania (7):
  - Bucharest
  - Craiova
  - Focşani
  - Oradea
  - Piteşti
  - Tg Mures
  - Timișoara
- Russia (32):
  - Arkhangelsk
  - Barnaul
  - Chelyabinsk
  - Ivanovo
  - Kaliningrad
  - Kemerovo
  - Kirov
  - Krasnodar
  - Krasnoyarsk
  - Kursk
  - Lyubertsy
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Orenburg
  - Penza
  - Perm
  - Pskov
  - Pushkin, Saint-Petersburg
  - Ryazan
  - Saint Petersburg
  - Saint-Petersbrug
  - Sestroretsk, Saint-Petersburg
  - Syktyvkar
  - Tomsk
  - Tula
  - Tumen Region
  - Vladimir
  - Voronezh
  - Yaroslavl Nap
  - Yekaterinburg
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Niška Banja
- Slovakia (3):
  - Bratislava
  - Nové Zámky
  - Žilina
- South Korea (5):
  - Daejeon
  - Gwangju
  - Seognam-Si, Kyungki-Do
  - Seoul
  - Suwon
- Spain (16):
  - Alicante
  - Aviles Asturias
  - Barcelona
  - Burgos
  - Elche
  - Figueres
  - Guadalajara
  - Huelva
  - Madrid
  - Málaga
  - Salamanca
  - Santander
  - Seville
  - Tarragona
  - Valencia
  - Vigo
- Sweden (9):
  - Danderyd
  - Gothenburg
  - Jönköping
  - Linköping
  - Lund
  - Malmo
  - Örebro
  - Östersund
  - Umeå
- Thailand (4):
  - Bangkok
  - Chiang Mai
  - Pathum Thani
  - Phathumwan
- Tunisia (3):
  - Sfax
  - Sousse
  - Tunis
- Turkey (Türkiye) (9):
  - Ankara
  - Aydin
  - Bursa
  - Erzurum
  - Istanbul
  - Izmir
  - Kayseri
  - Samsun
  - Sivas
- Ukraine (18):
  - Cherkassy
  - Dnipro
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Khemelnitskiy
  - Kiev
  - Luhansk
  - Lutsk
  - Lviv
  - Mykolayiv
  - Poltava
  - Sumy
  - Ternopil
  - Uzhhorod
  - Vinnitsa
  - Zaporizhzhya
  - Zhytomyr
- United Kingdom (18):
  - Birmingham
  - Blackpool
  - Bristol
  - Chertsey
  - Chesterfield
  - East Sussex
  - Exeter
  - Hampshire
  - Harrow
  - Hull
  - Leicester
  - Lincoln
  - Manchester
  - Middlesbrough
  - Portadown
  - Stockport
  - Warwick
  - Worcester

REFERENCES:
- [Derived] Chi G, AlKhalfan F, Lee JJ, Montazerin SM, Fitzgerald C, Korjian S, Omar W, Barnathan E, Plotnikov A, Gibson CM. Factors associated with early, late, and very late stent thrombosis among patients with acute coronary syndrome undergoing coronary stent placement: analysis from the ATLAS ACS 2-TIMI 51 trial. Front Cardiovasc Med. 2024 Jan 8;10:1269011. doi: 10.3389/fcvm.2023.1269011. eCollection 2023. PMID 38259304
- [Derived] Gibson WJ, Nafee T, Travis R, Yee M, Kerneis M, Ohman M, Gibson CM. Machine learning versus traditional risk stratification methods in acute coronary syndrome: a pooled randomized clinical trial analysis. J Thromb Thrombolysis. 2020 Jan;49(1):1-9. doi: 10.1007/s11239-019-01940-8. PMID 31535314
- [Derived] Gibson CM, Levitan B, Gibson WJ, Yee MK, Murphy SA, Yuan Z, Chakrabarti AK, Lee M, Braunwald E. Fatal or Irreversible Bleeding and Ischemic Events With Rivaroxaban in Acute Coronary Syndrome. J Am Coll Cardiol. 2018 Jul 10;72(2):129-136. doi: 10.1016/j.jacc.2018.04.055. PMID 29976285
- [Derived] Cavender MA, Gibson CM, Braunwald E, Wiviott SD, Murphy SA, Toda Kato E, Plotnikov AN, Amuchastegui M, Oude Ophuis T, van Hessen M, Mega JL. The effect of rivaroxaban on myocardial infarction in the ATLAS ACS 2 - TIMI 51 trial. Eur Heart J Acute Cardiovasc Care. 2015 Oct;4(5):468-74. doi: 10.1177/2048872614554109. Epub 2014 Oct 15. PMID 25318481
- [Derived] Gibson CM, Chakrabarti AK, Mega J, Bode C, Bassand JP, Verheugt FW, Bhatt DL, Goto S, Cohen M, Mohanavelu S, Burton P, Stone G, Braunwald E; ATLAS-ACS 2 TIMI 51 Investigators. Reduction of stent thrombosis in patients with acute coronary syndromes treated with rivaroxaban in ATLAS-ACS 2 TIMI 51. J Am Coll Cardiol. 2013 Jul 23;62(4):286-90. doi: 10.1016/j.jacc.2013.03.041. Epub 2013 Apr 16. PMID 23602776
- [Derived] Mega JL, Braunwald E, Murphy SA, Plotnikov AN, Burton P, Kiss RG, Parkhomenko A, Tendera M, Widimsky P, Gibson CM. Rivaroxaban in patients stabilized after a ST-segment elevation myocardial infarction: results from the ATLAS ACS-2-TIMI-51 trial (Anti-Xa Therapy to Lower Cardiovascular Events in Addition to Standard Therapy in Subjects with Acute Coronary Syndrome-Thrombolysis In Myocardial Infarction-51). J Am Coll Cardiol. 2013 May 7;61(18):1853-9. doi: 10.1016/j.jacc.2013.01.066. Epub 2013 Mar 7. PMID 23500262
- [Derived] Mega JL, Braunwald E, Wiviott SD, Bassand JP, Bhatt DL, Bode C, Burton P, Cohen M, Cook-Bruns N, Fox KA, Goto S, Murphy SA, Plotnikov AN, Schneider D, Sun X, Verheugt FW, Gibson CM; ATLAS ACS 2-TIMI 51 Investigators. Rivaroxaban in patients with a recent acute coronary syndrome. N Engl J Med. 2012 Jan 5;366(1):9-19. doi: 10.1056/NEJMoa1112277. Epub 2011 Nov 13. PMID 22077192
- [Derived] Gibson CM, Mega JL, Burton P, Goto S, Verheugt F, Bode C, Plotnikov A, Sun X, Cook-Bruns N, Braunwald E. Rationale and design of the Anti-Xa therapy to lower cardiovascular events in addition to standard therapy in subjects with acute coronary syndrome-thrombolysis in myocardial infarction 51 (ATLAS-ACS 2 TIMI 51) trial: a randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of rivaroxaban in subjects with acute coronary syndrome. Am Heart J. 2011 May;161(5):815-821.e6. doi: 10.1016/j.ahj.2011.01.026. PMID 21570509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study, an efficacy and safety study of rivaroxaban in patients with acute coronary syndrome, was conducted between 26 November 2008 and 19 September 2011. Patients were recruited from 766 study centers located in 44 countries worldwide.
Pre-assignment Details: A total of 15,526 patients were randomly allocated to the 3 treatment arms in the study. A total of 15,350 patients (5,115 patients in the rivaroxaban 2.5 mg bid group, 5,110 patients in the rivaroxaban 5 mg bid group and 5,125 patients in the placebo group) who received at least 1 dose of study drug were included in the safety analysis set.
Groups:
- Rivaroxaban 2.5 mg Bid: One rivaroxaban 2.5 mg tablet twice daily
- Rivaroxaban 5 mg Bid: One rivaroxaban 5 mg tablet twice daily
Period: Overall Study
Arm/Group | Placebo | Rivaroxaban 2.5 mg Bid | Rivaroxaban 5 mg Bid
Started | 5176 | 5174 | 5176
Treated/Safety Population | 5125 (All randomized participants who received at least one dose of study drug) | 5115 (All randomized participants who received at least one dose of study drug) | 5110 (All randomized participants who received at least one dose of study drug)
Modified Intent-to-Treat Population | 5113 (All randomized participants excluding 3 sites without regard to treatment exposure) | 5114 (All randomized participants excluding 3 sites without regard to treatment exposure) | 5115 (All randomized participants excluding 3 sites without regard to treatment exposure)
Completed | 4393 | 4399 | 4332
Not Completed | 783 | 775 | 844
Not completed — Death | 194 | 147 | 196
Not completed — Lost to Follow-up | 17 | 10 | 18
Not completed — Withdrawal by Subject | 405 | 448 | 441
Not completed — Other Reason | 167 | 170 | 189

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rivaroxaban 2.5 mg Bid | Rivaroxaban 5 mg Bid | Total
Number analyzed (Participants) | 5125 | 5115 | 5110 | 15350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3320 | 3239 | 3210 | 9769
  >=65 years | 1805 | 1876 | 1900 | 5581
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.38) | 61.8 (9.22) | 61.9 (9.00) | 61.7 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1280 | 1283 | 1316 | 3879
  Male | 3845 | 3832 | 3794 | 11471
Region of Enrollment [Number; unit: participants]
  Argentina | 118 | 126 | 158 | 402
  Australia | 172 | 182 | 150 | 504
  Belgium | 59 | 57 | 53 | 169
  Brazil | 184 | 171 | 168 | 523
  Bulgaria | 258 | 264 | 268 | 790
  Canada | 67 | 58 | 63 | 188
  Chile | 67 | 65 | 78 | 210
  China | 281 | 299 | 302 | 882
  Colombia | 97 | 84 | 87 | 268
  Croatia | 21 | 19 | 22 | 62
  Czech Republic | 154 | 158 | 170 | 482
  Denmark | 35 | 21 | 41 | 97
  Egypt | 63 | 47 | 46 | 156
  France | 68 | 67 | 72 | 207
  Germany | 101 | 96 | 122 | 319
  Greece | 19 | 21 | 27 | 67
  Hungary | 147 | 142 | 122 | 411
  India | 479 | 507 | 473 | 1459
  Israel | 114 | 122 | 101 | 337
  Italy | 78 | 77 | 77 | 232
  Japan | 131 | 135 | 131 | 397
  Latvia | 27 | 33 | 40 | 100
  Lithuania | 59 | 51 | 66 | 176
  Malaysia | 36 | 33 | 26 | 95
  Mexico | 71 | 96 | 86 | 253
  Morocco | 12 | 22 | 22 | 56
  Netherlands | 131 | 113 | 124 | 368
  New Zealand | 28 | 31 | 38 | 97
  Philippines | 19 | 11 | 8 | 38
  Poland | 332 | 361 | 356 | 1049
  Portugal | 36 | 36 | 43 | 115
  Romania | 103 | 94 | 107 | 304
  Russian Federation | 586 | 596 | 569 | 1751
  Serbia | 43 | 45 | 29 | 117
  Slovakia | 67 | 58 | 53 | 178
  South Korea | 57 | 40 | 49 | 146
  Spain | 71 | 73 | 76 | 220
  Sweden | 58 | 41 | 44 | 143
  Thailand | 52 | 50 | 38 | 140
  Tunisia | 60 | 62 | 52 | 174
  Turkey | 37 | 39 | 41 | 117
  Ukraine | 205 | 210 | 213 | 628
  United Kingdom | 79 | 91 | 75 | 245
  United States | 243 | 211 | 224 | 678

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With the Composite Endpoint of Cardiovascular Death, Myocardial Infarction, or Stroke
Description: The percentage of patients with the first occurrence of the composite of death, myocardial infarction, or stroke. The statistical analysis was based on the time from randomization to the first occurrence of the event while on treatment.
Time Frame: From the time of randomization (Day 1) up to completion of the treatment phase (Month 6)
Population: The Modified Intent-to-Treat (mITT) population consisted of all randomized patients, regardless of treatment exposure, excluding sites 091001, 091019, and 091026 (excluded due to potential trial misconduct). The mITT population was also subject to censoring of events that occurred on, or after, the global treatment end date.
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Rivaroxaban 2.5 mg Bid | Rivaroxaban 5 mg Bid
Number analyzed (Participants) | 5113 | 5114 | 5115
Percentage of patients | 7.4 | 6.1 | 6.1
Statistical Analysis 1: Comparison: Placebo vs Rivaroxaban 2.5 mg Bid; Test type: Superiority or Other; p = 0.020, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.72 to 0.97] — Based upon the Cox proportional hazards model
Statistical Analysis 2: Comparison: Placebo vs Rivaroxaban 5 mg Bid; Test type: Superiority or Other; p = 0.028, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.73 to 0.98] — Based upon the Cox proportional hazards model

2. Secondary Outcome: The Percentage of Patients With the Composite of All Cause Death, Myocardial Infarction, or Stroke
Description: The percentage of patients with the first occurrence of the composite endpoint. The statistical analysis was based on the time from randomization to the first occurrence of the event while on treatment.
Time Frame: From the time of randomization (Day 1) up to completion of the treatment phase (Month 6)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Rivaroxaban 2.5 mg Bid | Rivaroxaban 5 mg Bid
Number analyzed (Participants) | 5113 | 5114 | 5115
Percentage of patients | 7.5 | 6.3 | 6.3
Statistical Analysis 1: Comparison: Placebo vs Rivaroxaban 2.5 mg Bid; Test type: Superiority or Other; p = 0.016, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.72 to 0.97] — Based on the Cox proportional hazards model
Statistical Analysis 2: Comparison: Placebo vs Rivaroxaban 5 mg Bid; Test type: Superiority or Other; p = 0.025, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.73 to 0.98] — Based on the Cox proportional hazards model

3. Secondary Outcome: The Percentage of Patients With the Composite of Cardiovascular Death, Myocardial Infarction, Ischemic Stroke, or TIMI Major Bleeding Event Not Associated With Coronary Artery Bypass Graft Surgery
Description: as for outcome 2
Time Frame: From the time of randomization (Day 1) up to completion of the treatment phase (Month 6)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Rivaroxaban 2.5 mg Bid | Rivaroxaban 5 mg Bid
Number analyzed (Participants) | 5113 | 5114 | 5115
Percentage of patients | 7.6 | 7.1 | 7.2
Statistical Analysis 1: Comparison: Placebo vs Rivaroxaban 2.5 mg Bid; Test type: Superiority or Other; p = 0.320, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.81 to 1.07] — Based upon the Cox proportional hazards model
Statistical Analysis 2: Comparison: Placebo vs Rivaroxaban 5 mg Bid; Test type: Superiority or Other; p = 0.508, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.83 to 1.10] — Based upon the Cox proportional hazards model

4. Secondary Outcome: The Percentage of Patients With the Composite of Cardiovascular Death, Myocardial Infarction, Stroke, or Severe Recurrent Ischemia Requiring Revascularization
Description: as for outcome 2
Time Frame: From the time of randomization (Day 1) up to completion of the treatment phase (Month 6)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Rivaroxaban 2.5 mg Bid | Rivaroxaban 5 mg Bid
Number analyzed (Participants) | 5113 | 5114 | 5115
Percentage of patients | 9.4 | 8.5 | 8.2
Statistical Analysis 1: Comparison: Placebo vs Rivaroxaban 2.5 mg Bid; Test type: Superiority or Other; p = 0.185, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.80 to 1.04] — Based upon the Cox proportional hazards model
Statistical Analysis 2: Comparison: Placebo vs Rivaroxaban 5 mg Bid; Test type: Superiority or Other; p = 0.081, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.78 to 1.01] — Based upon the Cox proportional hazards model

5. Secondary Outcome: The Percentage of Patients With the Composite of Cardiovascular Death, Myocardial Infarction, Stroke, or Severe Recurrent Ischemia Leading to Hospitalization
Description: as for outcome 2
Time Frame: From the time of randomization (Day 1) up to completion of the treatment phase (Month 6)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Rivaroxaban 2.5 mg Bid | Rivaroxaban 5 mg Bid
Number analyzed (Participants) | 5113 | 5114 | 5115
Percentage of patients | 8.7 | 7.3 | 7.6
Statistical Analysis 1: Comparison: Placebo vs Rivaroxaban 2.5 mg Bid; Test type: Superiority or Other; p = 0.011, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.73 to 0.96] — Based upon the Cox proportional hazards model
Statistical Analysis 2: Comparison: Placebo vs Rivaroxaban 5 mg Bid; Test type: Superiority or Other; p = 0.070, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.78 to 1.01] — Based upon the Cox proportional hazards model

ADVERSE EVENTS:
Arm/Group | Placebo | Rivaroxaban 2.5 mg Bid | Rivaroxaban 5 mg Bid
Serious Adverse Events (participants affected / at risk) | 1018/5125 | 1033/5115 | 1083/5110
Other Adverse Events (participants affected / at risk) | 140/5125 | 259/5115 | 341/5110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5125) | Rivaroxaban 2.5 mg Bid (N=5115) | Rivaroxaban 5 mg Bid (N=5110)
Anaemia (Blood and lymphatic system disorders) | 3 | 6 | 11
Anaemia Megaloblastic (Blood and lymphatic system disorders) | 0 | 0 | 1
Aplastic Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Spontaneous Haematoma (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 9 | 7 | 7
Acute Left Ventricular Failure (Cardiac disorders) | 2 | 4 | 3
Acute Myocardial Infarction (Cardiac disorders) | 25 | 15 | 17
Adams-Stokes Syndrome (Cardiac disorders) | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 118 | 93 | 106
Angina Unstable (Cardiac disorders) | 100 | 105 | 123
Aortic Valve Disease (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 4 | 1 | 4
Arrhythmia Supraventricular (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 27 | 27 | 21
Atrial Flutter (Cardiac disorders) | 4 | 3 | 8
Atrial Tachycardia (Cardiac disorders) | 1 | 0 | 1
Atrioventricular Block (Cardiac disorders) | 2 | 0 | 0
Atrioventricular Block Complete (Cardiac disorders) | 2 | 5 | 4
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 3 | 1
Bradycardia (Cardiac disorders) | 1 | 1 | 3
Bundle Branch Block Left (Cardiac disorders) | 0 | 0 | 1
Bundle Branch Block Right (Cardiac disorders) | 0 | 0 | 1
Cardiac Aneurysm (Cardiac disorders) | 0 | 0 | 2
Cardiac Arrest (Cardiac disorders) | 9 | 5 | 7
Cardiac Asthma (Cardiac disorders) | 0 | 1 | 1
Cardiac Failure (Cardiac disorders) | 41 | 56 | 27
Cardiac Failure Acute (Cardiac disorders) | 13 | 14 | 10
Cardiac Failure Chronic (Cardiac disorders) | 4 | 6 | 7
Cardiac Failure Congestive (Cardiac disorders) | 21 | 15 | 20
Cardiac Flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac Pseudoaneurysm (Cardiac disorders) | 0 | 1 | 1
Cardiac Tamponade (Cardiac disorders) | 1 | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 2 | 2
Cardiogenic Shock (Cardiac disorders) | 7 | 9 | 4
Cardiovascular Insufficiency (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Aneurysm (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 16 | 26 | 13
Coronary Artery Dissection (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Insufficiency (Cardiac disorders) | 2 | 0 | 0
Coronary Artery Stenosis (Cardiac disorders) | 3 | 3 | 7
Dressler's Syndrome (Cardiac disorders) | 1 | 1 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 2
Intracardiac Thrombus (Cardiac disorders) | 3 | 0 | 2
Ischaemic Cardiomyopathy (Cardiac disorders) | 2 | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 2 | 2 | 2
Left Ventricular Failure (Cardiac disorders) | 6 | 7 | 5
Mitral Valve Incompetence (Cardiac disorders) | 0 | 2 | 0
Myocardial Infarction (Cardiac disorders) | 16 | 10 | 22
Myocardial Ischaemia (Cardiac disorders) | 13 | 15 | 15
Myocardial Rupture (Cardiac disorders) | 3 | 0 | 1
Nodal Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Nodal Rhythm (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 2 | 3
Papillary Muscle Rupture (Cardiac disorders) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 1
Pericardial Haemorrhage (Cardiac disorders) | 0 | 0 | 4
Pericarditis (Cardiac disorders) | 1 | 1 | 2
Postinfarction Angina (Cardiac disorders) | 2 | 0 | 1
Prinzmetal Angina (Cardiac disorders) | 1 | 0 | 0
Right Ventricular Failure (Cardiac disorders) | 1 | 0 | 0
Sick Sinus Syndrome (Cardiac disorders) | 2 | 3 | 0
Silent Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Sinoatrial Block (Cardiac disorders) | 1 | 1 | 1
Sinus Arrhythmia (Cardiac disorders) | 2 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 2 | 3 | 6
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 2 | 0
Tachycardia Paroxysmal (Cardiac disorders) | 1 | 0 | 0
Torsade De Pointes (Cardiac disorders) | 1 | 0 | 0
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 1 | 1 | 1
Ventricular Fibrillation (Cardiac disorders) | 8 | 6 | 8
Ventricular Tachycardia (Cardiac disorders) | 10 | 10 | 4
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 | 0 | 0
Gastrointestinal Angiodysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Hip Dysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0
Acute Vestibular Syndrome (Ear and labyrinth disorders) | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 1 | 0 | 1
Ear Haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 1
Middle Ear Inflammation (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 3 | 3
Vertigo Positional (Ear and labyrinth disorders) | 0 | 1 | 0
Autoimmune Thyroiditis (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 5 | 3 | 1
Conjunctival Haemorrhage (Eye disorders) | 1 | 0 | 0
Eye Haemorrhage (Eye disorders) | 3 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Hyphaema (Eye disorders) | 0 | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1 | 0
Vitreous Haemorrhage (Eye disorders) | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 5 | 5 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 4 | 3
Anal Fissure (Gastrointestinal disorders) | 1 | 2 | 2
Anal Fistula (Gastrointestinal disorders) | 1 | 0 | 1
Appendix Disorder (Gastrointestinal disorders) | 0 | 1 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Colonic Polyp (Gastrointestinal disorders) | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 3
Diverticulitis Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 2 | 1 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Erosive Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 1 | 0
Gastric Dysplasia (Gastrointestinal disorders) | 1 | 0 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 2 | 2 | 3
Gastric Polyps (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 4 | 2 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 3 | 0
Gastritis (Gastrointestinal disorders) | 7 | 5 | 4
Gastritis Erosive (Gastrointestinal disorders) | 0 | 3 | 6
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 11 | 18 | 32
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 1 | 1
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0 | 2
Gingival Swelling (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 4
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhagic Erosive Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 4 | 8
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 3
Ileus (Gastrointestinal disorders) | 1 | 1 | 1
Ileus Paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 2 | 2 | 5
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 3
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 2
Intestinal Polyp Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 3
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 4 | 7 | 8
Mesenteric Panniculitis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Oesophageal Spasm (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 1 | 0
Pancreatic Necrosis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 6 | 4 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 3 | 6 | 2
Pancreatitis Chronic (Gastrointestinal disorders) | 2 | 2 | 1
Peptic Ulcer (Gastrointestinal disorders) | 0 | 2 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 1
Periproctitis (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 2 | 0
Proctocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Pseudodiverticular Disease (Gastrointestinal disorders) | 0 | 0 | 1
Radicular Cyst (Gastrointestinal disorders) | 0 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 4 | 9 | 8
Rectal Polyp (Gastrointestinal disorders) | 0 | 2 | 0
Reflux Oesophagitis (Gastrointestinal disorders) | 2 | 1 | 0
Retroperitoneal Haematoma (Gastrointestinal disorders) | 0 | 1 | 1
Salivary Gland Cyst (Gastrointestinal disorders) | 1 | 0 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 2 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 5 | 9 | 14
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0
Accidental Death (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 2 | 0 | 1
Cardiac Death (General disorders) | 1 | 0 | 1
Chest Discomfort (General disorders) | 1 | 2 | 3
Chest Pain (General disorders) | 33 | 47 | 33
Condition Aggravated (General disorders) | 0 | 0 | 1
Cyst Rupture (General disorders) | 0 | 0 | 1
Death (General disorders) | 11 | 5 | 9
Device Lead Damage (General disorders) | 1 | 0 | 0
Device Occlusion (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 2
Gait Disturbance (General disorders) | 0 | 1 | 1
Generalised Oedema (General disorders) | 1 | 0 | 0
Hernia (General disorders) | 0 | 1 | 0
Hernia Obstructive (General disorders) | 0 | 0 | 1
Impaired Healing (General disorders) | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Medical Device Complication (General disorders) | 1 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 39 | 36 | 48
Oedema Peripheral (General disorders) | 0 | 1 | 0
Puncture Site Haemorrhage (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 5 | 7
Sudden Cardiac Death (General disorders) | 13 | 9 | 10
Sudden Death (General disorders) | 36 | 23 | 29
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 0 | 1
Thrombosis in Device (General disorders) | 2 | 1 | 2
Vessel Puncture Site Haematoma (General disorders) | 0 | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 1 | 2
Biliary Colic (Hepatobiliary disorders) | 0 | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 7 | 8 | 9
Cholecystitis Acute (Hepatobiliary disorders) | 3 | 4 | 2
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 4 | 3 | 4
Hepatic Failure (Hepatobiliary disorders) | 2 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 2 | 2
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 2
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 1 | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Immune Reconstitution Syndrome (Immune system disorders) | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 1
Anal Abscess (Infections and infestations) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 3 | 1 | 3
Appendicitis Perforated (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 1
Bacterial Prostatitis (Infections and infestations) | 0 | 1 | 0
Borrelia Infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 5 | 5
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 5 | 7 | 1
Clostridial Infection (Infections and infestations) | 1 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Dengue Fever (Infections and infestations) | 0 | 2 | 0
Device Related Infection (Infections and infestations) | 1 | 0 | 0
Diabetic Gangrene (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 3 | 0 | 0
Empyema (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Enteritis Infectious (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Eyelid Infection (Infections and infestations) | 0 | 0 | 1
Gangrene (Infections and infestations) | 1 | 2 | 1
Gastroenteritis (Infections and infestations) | 4 | 6 | 4
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 1 | 0 | 0
Graft Infection (Infections and infestations) | 0 | 1 | 0
Groin Abscess (Infections and infestations) | 0 | 1 | 0
Groin Infection (Infections and infestations) | 0 | 0 | 1
H1n1 Influenza (Infections and infestations) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Hepatitis E (Infections and infestations) | 1 | 0 | 1
Hepatitis Viral (Infections and infestations) | 1 | 1 | 0
Herpes Zoster (Infections and infestations) | 2 | 1 | 2
Herpes Zoster Infection Neurological (Infections and infestations) | 1 | 0 | 0
Incision Site Infection (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 1
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 0 | 1 | 1
Infective Spondylitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Localised Infection (Infections and infestations) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 2 | 0
Lung Abscess (Infections and infestations) | 0 | 1 | 0
Lung Infection (Infections and infestations) | 2 | 3 | 1
Lymphangitis (Infections and infestations) | 0 | 1 | 0
Mediastinitis (Infections and infestations) | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 1 | 1
Meningitis Pneumococcal (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Neutropenic Infection (Infections and infestations) | 0 | 1 | 0
Oesophageal Candidiasis (Infections and infestations) | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Otitis Externa (Infections and infestations) | 0 | 0 | 1
Otitis Media Chronic (Infections and infestations) | 1 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Pericoronitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 33 | 37 | 33
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia Viral (Infections and infestations) | 0 | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 2 | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 2 | 2 | 0
Pyelonephritis Chronic (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 5 | 1 | 3
Septic Shock (Infections and infestations) | 1 | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Skin Infection (Infections and infestations) | 1 | 0 | 1
Staphylococcal Abscess (Infections and infestations) | 2 | 0 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1 | 2
Tinea Pedis (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 2 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 8 | 9 | 9
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 1 | 1
Urosepsis (Infections and infestations) | 2 | 2 | 5
Vestibular Neuronitis (Infections and infestations) | 0 | 0 | 1
Viral Infection (Infections and infestations) | 2 | 0 | 1
Viral Myocarditis (Infections and infestations) | 0 | 0 | 1
Wound Infection (Infections and infestations) | 3 | 2 | 0
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Airway Burns (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anaphylactic Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anastomotic Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anastomotic Ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 1
Animal Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Brain Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Cardiac Procedure Complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Cerebral Haemorrhage Traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0
Chemical Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 2 | 2
Contrast Media Reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 0 | 5 | 2
Extradural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 | 2 | 2
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 3
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured Skull Depressed (Injury, poisoning and procedural complications) | 0 | 1 | 0
Haematuria Traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 3 | 3 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
In-Stent Arterial Restenosis (Injury, poisoning and procedural complications) | 1 | 1 | 2
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 4 | 3 | 7
Incision Site Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 2 | 1
Muscle Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Operative Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 5 | 3 | 5
Post Procedural Myocardial Infarction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural Site Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Renal Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 3 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 3 | 2
Spinal Column Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic Rupture (Injury, poisoning and procedural complications) | 2 | 1 | 2
Stab Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sternal Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 3
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 | 1 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Traumatic Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 3 | 8 | 5
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound Necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 21 | 24 | 21
Angiogram (Investigations) | 0 | 1 | 0
Arteriogram Coronary (Investigations) | 5 | 4 | 6
Aspartate Aminotransferase Increased (Investigations) | 1 | 1 | 1
Blood Bilirubin Increased (Investigations) | 0 | 2 | 0
Blood Creatinine Increased (Investigations) | 0 | 2 | 2
Blood Glucose Increased (Investigations) | 1 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 1 | 3
Cardiac Stress Test (Investigations) | 0 | 1 | 0
Cardiac Stress Test Abnormal (Investigations) | 1 | 1 | 0
Colonoscopy (Investigations) | 0 | 1 | 0
Ejection Fraction Decreased (Investigations) | 1 | 0 | 0
Electrocardiogram Change (Investigations) | 0 | 0 | 1
Electrocardiogram St-T Change (Investigations) | 1 | 0 | 0
Endoscopy Upper Gastrointestinal Tract (Investigations) | 0 | 0 | 2
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 1 | 1
Haemoglobin Decreased (Investigations) | 1 | 8 | 5
Hepatic Enzyme Increased (Investigations) | 4 | 7 | 7
Liver Function Test Abnormal (Investigations) | 5 | 6 | 6
Occult Blood Positive (Investigations) | 0 | 1 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 1
Renal Function Test Abnormal (Investigations) | 1 | 0 | 0
Transaminases Increased (Investigations) | 2 | 0 | 0
Troponin I Increased (Investigations) | 0 | 1 | 0
Ultrasound Scan (Investigations) | 1 | 0 | 0
Weight Decreased (Investigations) | 2 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 9 | 12 | 9
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2 | 1 | 1
Diabetic Foot (Metabolism and nutrition disorders) | 1 | 1 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 2 | 1
Fluid Overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Bone Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral Disc Displacement (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1
Jaw Cyst (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adrenal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 2
Breast Cancer Female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0
Cardiac Myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ear Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Female Reproductive Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 2
Gastric Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Laryngeal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 3
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mesothelioma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastatic Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oropharyngeal Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Polycythaemia Vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 5
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Rectal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Salivary Gland Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Signet-Ring Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous Cell Carcinoma of the Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Urinary Tract Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Vaginal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1
Basal Ganglia Haemorrhage (Nervous system disorders) | 0 | 1 | 0
Brain Injury (Nervous system disorders) | 0 | 1 | 0
Brain Oedema (Nervous system disorders) | 0 | 1 | 0
Brain Stem Infarction (Nervous system disorders) | 0 | 1 | 0
Carotid Arteriosclerosis (Nervous system disorders) | 0 | 1 | 0
Carotid Artery Disease (Nervous system disorders) | 0 | 1 | 0
Carotid Artery Occlusion (Nervous system disorders) | 0 | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 2 | 0
Cerebellar Haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral Artery Embolism (Nervous system disorders) | 0 | 0 | 2
Cerebral Artery Stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 3 | 1 | 4
Cerebral Infarction (Nervous system disorders) | 2 | 1 | 5
Cerebrovascular Accident (Nervous system disorders) | 2 | 5 | 5
Cerebrovascular Disorder (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Insufficiency (Nervous system disorders) | 1 | 0 | 0
Coma (Nervous system disorders) | 0 | 1 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 2
Diabetic Neuropathy (Nervous system disorders) | 2 | 3 | 0
Dizziness (Nervous system disorders) | 6 | 5 | 4
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 1 | 0
Grand Mal Convulsion (Nervous system disorders) | 0 | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 0 | 6 | 9
Haemorrhagic Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic Stroke (Nervous system disorders) | 3 | 1 | 3
Headache (Nervous system disorders) | 1 | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hypertensive Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Intercostal Neuralgia (Nervous system disorders) | 0 | 1 | 0
Intracranial Haematoma (Nervous system disorders) | 0 | 1 | 0
Intraventricular Haemorrhage (Nervous system disorders) | 0 | 0 | 1
Ischaemic Cerebral Infarction (Nervous system disorders) | 5 | 2 | 4
Ischaemic Stroke (Nervous system disorders) | 18 | 12 | 16
Lacunar Infarction (Nervous system disorders) | 6 | 4 | 0
Loss of Consciousness (Nervous system disorders) | 2 | 2 | 2
Lumbar Radiculopathy (Nervous system disorders) | 1 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Peripheral Nerve Palsy (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 2 | 3
Radiculitis Cervical (Nervous system disorders) | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Speech Disorder (Nervous system disorders) | 1 | 0 | 1
Spinal Claudication (Nervous system disorders) | 1 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 1 | 3
Syncope (Nervous system disorders) | 11 | 6 | 16
Thalamus Haemorrhage (Nervous system disorders) | 0 | 1 | 0
Thrombotic Cerebral Infarction (Nervous system disorders) | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 10 | 4 | 10
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 | 1 | 1
Viith Nerve Paralysis (Nervous system disorders) | 0 | 1 | 1
Acute Psychosis (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 1 | 1
Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 0
Burnout Syndrome (Psychiatric disorders) | 0 | 0 | 1
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
Major Depression (Psychiatric disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 1
Neurosis (Psychiatric disorders) | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
Bladder Disorder (Renal and urinary disorders) | 0 | 0 | 1
Bladder Obstruction (Renal and urinary disorders) | 1 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 0 | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 3 | 2 | 1
Diabetic Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 7 | 21
Haemorrhage Urinary Tract (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1
Hypertensive Nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 3 | 3
Neurogenic Bladder (Renal and urinary disorders) | 1 | 0 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 1 | 2 | 0
Renal Colic (Renal and urinary disorders) | 1 | 1 | 3
Renal Failure (Renal and urinary disorders) | 4 | 2 | 0
Renal Failure Acute (Renal and urinary disorders) | 3 | 3 | 2
Renal Failure Chronic (Renal and urinary disorders) | 0 | 0 | 2
Renal Haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 2 | 1 | 0
Renal Mass (Renal and urinary disorders) | 1 | 0 | 0
Urethral Haemorrhage (Renal and urinary disorders) | 0 | 2 | 0
Urethral Meatus Stenosis (Renal and urinary disorders) | 0 | 0 | 1
Urinary Bladder Polyp (Renal and urinary disorders) | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 3 | 1 | 4
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 2 | 1 | 4
Calculus Prostatic (Reproductive system and breast disorders) | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 2
Leukoplakia of Penis (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 2
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 1 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 4 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 6
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Brain Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchial Fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 12 | 11
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Dyspnoea at Rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 10 | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 11
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Henoch-Schonlein Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cardiac Valve Prosthesis User (Social circumstances) | 1 | 0 | 0
Prosthesis User (Social circumstances) | 1 | 0 | 0
Angioplasty (Surgical and medical procedures) | 0 | 3 | 0
Aortic Aneurysm Repair (Surgical and medical procedures) | 0 | 0 | 1
Aortic Valve Replacement (Surgical and medical procedures) | 0 | 1 | 0
Arterial Repair (Surgical and medical procedures) | 0 | 1 | 0
Arteriovenous Shunt Operation (Surgical and medical procedures) | 0 | 0 | 1
Bladder Neoplasm Surgery (Surgical and medical procedures) | 0 | 0 | 1
Cardiac Ablation (Surgical and medical procedures) | 0 | 1 | 0
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 1 | 1 | 0
Carotid Endarterectomy (Surgical and medical procedures) | 0 | 1 | 1
Cataract Operation (Surgical and medical procedures) | 1 | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 2 | 2
Coronary Angioplasty (Surgical and medical procedures) | 0 | 1 | 1
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 0 | 0 | 1
Coronary Artery Bypass (Surgical and medical procedures) | 3 | 3 | 6
Coronary Revascularisation (Surgical and medical procedures) | 2 | 1 | 1
Foot Amputation (Surgical and medical procedures) | 1 | 0 | 0
Gastric Banding (Surgical and medical procedures) | 1 | 0 | 0
Gastric Bypass (Surgical and medical procedures) | 1 | 0 | 0
Glaucoma Surgery (Surgical and medical procedures) | 0 | 1 | 0
Hernia Repair (Surgical and medical procedures) | 0 | 1 | 0
Hip Arthroplasty (Surgical and medical procedures) | 2 | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 1
Implantable Defibrillator Insertion (Surgical and medical procedures) | 0 | 1 | 2
Inguinal Hernia Repair (Surgical and medical procedures) | 1 | 1 | 1
Knee Arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Knee Operation (Surgical and medical procedures) | 1 | 2 | 0
Leg Amputation (Surgical and medical procedures) | 1 | 0 | 0
Meniscus Operation (Surgical and medical procedures) | 0 | 0 | 1
Orthopedic Procedure (Surgical and medical procedures) | 1 | 0 | 0
Pancreas Transplant (Surgical and medical procedures) | 1 | 0 | 0
Percutaneous Coronary Intervention (Surgical and medical procedures) | 5 | 10 | 8
Polypectomy (Surgical and medical procedures) | 0 | 1 | 1
Prostatectomy (Surgical and medical procedures) | 1 | 0 | 0
Rehabilitation Therapy (Surgical and medical procedures) | 2 | 0 | 0
Shoulder Operation (Surgical and medical procedures) | 0 | 0 | 1
Spinal Laminectomy (Surgical and medical procedures) | 0 | 1 | 0
Thyroidectomy (Surgical and medical procedures) | 0 | 1 | 0
Tooth Extraction (Surgical and medical procedures) | 0 | 0 | 1
Tracheostomy Tube Removal (Surgical and medical procedures) | 0 | 1 | 0
Transurethral Prostatectomy (Surgical and medical procedures) | 0 | 1 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 1 | 0
Angiopathy (Vascular disorders) | 0 | 1 | 0
Aortic Aneurysm (Vascular disorders) | 4 | 2 | 2
Aortic Dissection (Vascular disorders) | 1 | 0 | 0
Aortic Stenosis (Vascular disorders) | 0 | 1 | 1
Arterial Disorder (Vascular disorders) | 0 | 1 | 1
Arterial Thrombosis (Vascular disorders) | 0 | 0 | 1
Arterial Thrombosis Limb (Vascular disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 2 | 1 | 0
Arteriosclerosis Obliterans (Vascular disorders) | 2 | 1 | 2
Arteriovenous Fistula (Vascular disorders) | 1 | 0 | 1
Arteritis (Vascular disorders) | 0 | 0 | 1
Artery Dissection (Vascular disorders) | 0 | 1 | 0
Blue Toe Syndrome (Vascular disorders) | 0 | 1 | 0
Circulatory Collapse (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1 | 1
Diabetic Vascular Disorder (Vascular disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 1
Extremity Necrosis (Vascular disorders) | 1 | 0 | 0
Femoral Arterial Stenosis (Vascular disorders) | 2 | 0 | 0
Femoral Artery Embolism (Vascular disorders) | 1 | 0 | 0
Femoral Artery Occlusion (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 2 | 7 | 6
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 8 | 16 | 6
Hypertensive Crisis (Vascular disorders) | 10 | 8 | 14
Hypertensive Emergency (Vascular disorders) | 3 | 0 | 2
Hypotension (Vascular disorders) | 3 | 5 | 5
Hypovolaemic Shock (Vascular disorders) | 1 | 1 | 0
Iliac Artery Occlusion (Vascular disorders) | 1 | 0 | 0
Intermittent Claudication (Vascular disorders) | 3 | 1 | 3
Intra-Abdominal Haemorrhage (Vascular disorders) | 0 | 0 | 1
Ischaemia (Vascular disorders) | 2 | 0 | 0
Leriche Syndrome (Vascular disorders) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 2
Peripheral Arterial Occlusive Disease (Vascular disorders) | 4 | 3 | 5
Peripheral Artery Aneurysm (Vascular disorders) | 1 | 0 | 2
Peripheral Embolism (Vascular disorders) | 1 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0 | 1
Peripheral Vascular Disorder (Vascular disorders) | 3 | 2 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 2 | 0
Thrombosis (Vascular disorders) | 1 | 2 | 0
Varicose Vein (Vascular disorders) | 1 | 0 | 0
Vasospasm (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5125) | Rivaroxaban 2.5 mg Bid (N=5115) | Rivaroxaban 5 mg Bid (N=5110)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 140 | 259 | 341

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.